CLINICAL TRIAL: NCT07035821
Title: Olanzapine for the Treatment of Breakthrough Chemotherapy-Induced Vomiting in Children: An Open-label, Randomized Phase 3 Trial
Brief Title: Olanzapine for Prevention of Vomiting in Children and Adolescents Receiving Highly Emetogenic Chemotherapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: scmc
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breakthrough Chemotherapy-Induced Vomiting (CIV) in Pediatric Patients; Pediatric Cancer
Keywords: chemotherapy; olanzapine; pediatric cancer; vomiting
MeSH Terms: conditions — Neoplasms; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Intervention Model Description: The control group gave patients oral placebo, while the experimental group gave patients oral olanzapine
Who Masked: Participant, Care Provider
Masking Description: Patients were randomized to one of the prespecified two arms (arm A: olanzapine or arm B: placebo) if they developed breakthrough vomiting. The department of biostatistics and cancer registry at the institute assisted in the random allocation of the patients. Randomization was performed by generating random number tables through customized computer program or the proposed total number of cases in the study, and the randomization codes were kept in sequentially numbered sealed envelopes. The envelopes were kept in the pediatric ward and opened when a patient was identified for randomization. A document was then prepared giving the allocation of all the subjects to the two arms in chronological order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olanzapine group (Experimental): Oral olanzapine tablets
  Interventions: Drug: Olanzapine Tablets
- Control group (Placebo Comparator): Oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine Tablets — Oral olanzapine tablets
  Arms: Olanzapine group
Drug: Placebo — Oral placebo
  Arms: Control group

SUMMARY:
Breakthrough chemotherapy-induced vomiting (CIV) is defined as CIV occurring after adequate antiemetic prophylaxis. Olanzapine is recommended for the treatment of breakthrough CIV in children, without adequate evidence. We conducted an open-label, single-center, phase 3 randomized controlled trial comparing the safety and efficacy of olanzapine and metoclopramide for treating breakthrough CIV.

DETAILED DESCRIPTION:
Children aged 5-18 years who developed breakthrough CIV after receiving highly emetogenic chemotherapy were randomly assigned to the control(placebo) or olanzapine arm. The primary objective of the study was to compare the complete response (CR) rates between patients receiving olanzapine or placebo for treating breakthrough CIV during 72 hours after the administration of the study drug. Secondary objectives were to compare CR rates for nausea and toxicities between the two arms.

ELIGIBILITY:
Inclusion Criteria:

- The major inclusion criteria were children aged 5 to 18 years at the time of study entry with documented cancer; receiving NK-1 inhibitor (aprepitant/fosaprepitant) and 5HT-3 antagonist (ondansetron) and/or dexamethasone as prophylactic antiemetics for CINV due to MEC or HEC; minimum body weight of 10 kg; development of breakthrough vomiting after starting prophylactic antiemetics; Lansky performance scale of above 50 (for patients aged 10 years or less) or Eastern Cooperative Oncology Group performance scale less than 3 and normal electrocardiogram (ECG) before the initiation of the prophylactic antiemetics.

Exclusion Criteria:

* Children with history of allergy to olanzapine or metoclopramide; patient with renal failure, congestive heart failure, or any uncontrolled disease except for malignancy; serum creatinine more than upper limit of normal (ULN) for age; serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) four times the ULN for age and serum bilirubin 1.5 times ULN for age; patient with history of central nervous system disease including brain metastasis, seizure disorder, or psychosis; patients on treatment with other antipsychotic agents such as risperidone, quetiapine, clozapine, or phenothiazine.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
the CR rate for vomiting in the first 72 hours | in the first 72 hours of the initiation of olanzapine
  The primary endpoint was the CR rate for vomiting in the first 72 hours of the initiation of olanzapine .

SECONDARY OUTCOMES:
the CR rate for nausea in the first 72 hours of the initiation of olanzapine | in the first 72 hours of the initiation of olanzapine
  The secondary endpoint was the CR rate for nausea in the first 72 hours of the initiation of olanzapine

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radhakrishnan V, Pai V, Rajaraman S, Mehra N, Ganesan T, Dhanushkodi M, Perumal Kalaiyarasi J, Rajan AK, Selvarajan G, Ranganathan R, Karunakaran P, Sagar TG. Olanzapine versus metoclopramide for the treatment of breakthrough chemotherapy-induced vomiting in children: An open-label, randomized phase 3 trial. Pediatr Blood Cancer. 2020 Sep;67(9):e28532. doi: 10.1002/pbc.28532. Epub 2020 Jun 22. PMID 32568452
- [Background] Moshayedi M, Salehifar E, Karami H, Hendouei N, Mousazadeh M, Alizadeh Haji S. Efficacy and Safety of Adding Olanzapine to the Standard Preventive Regimen for Chemotherapy-induced Nausea and Vomiting in Children: A Randomized Double-blind Controlled Trial. Iran J Pharm Res. 2021 Winter;20(1):318-326. doi: 10.22037/ijpr.2019.112514.13803. PMID 34400961
- [Background] Meena JP, Gupta AK, Jat KR, Anandani G, Sasidharan A, Tanwar P. Efficacy and Safety of Olanzapine for the Prevention of Chemotherapy-induced Nausea and Vomiting in Children: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Pediatr Hematol Oncol. 2023 Oct 1;45(7):361-369. doi: 10.1097/MPH.0000000000002737. Epub 2023 Aug 3. PMID 37539996
- [Background] Yoodee J, Permsuwan U, Nimworapan M. Efficacy and safety of olanzapine for the prevention of chemotherapy-induced nausea and vomiting: A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2017 Apr;112:113-125. doi: 10.1016/j.critrevonc.2017.02.017. Epub 2017 Feb 20. PMID 28325253
- [Background] Chiu L, Chow R, Popovic M, Navari RM, Shumway NM, Chiu N, Lam H, Milakovic M, Pasetka M, Vuong S, Chow E, DeAngelis C. Efficacy of olanzapine for the prophylaxis and rescue of chemotherapy-induced nausea and vomiting (CINV): a systematic review and meta-analysis. Support Care Cancer. 2016 May;24(5):2381-2392. doi: 10.1007/s00520-016-3075-8. Epub 2016 Jan 15. PMID 26768437
- [Background] Naik RD, V S, Singh V, Pillai AS, Dhawan D, Bakhshi S. Olanzapine for Prevention of Vomiting in Children and Adolescents Receiving Highly Emetogenic Chemotherapy: Investigator-Initiated, Randomized, Open-Label Trial. J Clin Oncol. 2020 Nov 10;38(32):3785-3793. doi: 10.1200/JCO.20.00871. Epub 2020 Sep 15. PMID 32931400
- [Background] Sutherland A, Naessens K, Plugge E, Ware L, Head K, Burton MJ, Wee B. Olanzapine for the prevention and treatment of cancer-related nausea and vomiting in adults. Cochrane Database Syst Rev. 2018 Sep 21;9(9):CD012555. doi: 10.1002/14651858.CD012555.pub2. PMID 30246876